CLINICAL TRIAL: NCT04168684
Title: Intervening Early With Neglected Children: Key Adolescent Outcomes
Brief Title: Intervening Early: Key Adolescent Outcomes
Acronym: SCOH-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Delaware (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIMH074374adol; R01MH074374 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-11-19 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Depressive Symptoms; Conduct Disorder; Anxiety Disorders
MeSH Terms: conditions — Depression; Conduct Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Families randomized to Attachment and Biobehavioral Catch-up (ABC) or to a control intervention (DEF)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parents received an intervention but did not know whether it was experimental or control. All participants had an identification number that did not indicate group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attachment and Biobehavioral Catch-up (ABC) (Experimental): 10 sessions that focused on parental nurturance, and sensitivity
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC)
- Developmental Education for Families (DEF) (Active Comparator): 10 sessions that focused on cognitive development
  Interventions: Behavioral: Developmental Education for Families (DEF)

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up (ABC) — Manualized intervention implemented in home with parent and child present focused on parental responsiveness
  Arms: Attachment and Biobehavioral Catch-up (ABC)
Behavioral: Developmental Education for Families (DEF) — Manualized intervention implemented in home with parent and child present focused on parental enhancement of child learning
  Arms: Developmental Education for Families (DEF)

SUMMARY:
This study follows children into adolescence who were first randomized to intervention condition in infancy.

DETAILED DESCRIPTION:
Parents serve as co-regulators for their young children, helping them regulate behaviors, emotions, and physiology and supporting the development of healthy brain circuitry. Neglecting parents often fail to serve as co-regulators, which has implications for young children's self-regulatory capabilities and brain development. As children become older, these difficulties with self-regulation may become more pronounced. Adolescence represents a period of particular vulnerability for the emergence of mental health problems because of increasing demands for regulation of emotions and behaviors, coupled with on-going development of neural circuits that support emotional and behavioral regulation. The Attachment and Biobehavioral Catch-up (ABC) intervention was designed to help parents learn to interact in responsive and sensitive ways, with the expectation that children would show enhanced ability to regulate behavior, emotions, and physiology. The efficacy of the ABC intervention among parents involved with Child Protective Services (CPS) was assessed. Parents were randomized to ABC or to a control intervention. Children were followed at T1 (ages 1-4) and T2 (ages 8-10). At T1, more of the children in the ABC group developed secure and organized attachments than children in the DEF group, and children in ABC showed more normative production of cortisol, less expression of negative emotions, and poorer inhibitory control than children in DEF. ABC parents were more sensitive and showed more optimal neural activity than DEF parents. At T2, ABC children showed greater prefrontal cortex activation in response to threat than DEF children, suggesting better regulation to threat at the level of brain activation. Also at T2, children in the ABC group reported more secure relationships with parents, and showed more normative cortisol production and more optimal autonomic nervous system functioning than DEF children. In adolescence, the ABC intervention is expected to result in enhanced brain circuitry and more optimal functioning across domains as assessed at multiple levels of analysis relative to the control intervention. In the proposed study, behavioral and neurobiological development among 13-, 14- and 15-year-old adolescents whose parents were referred by CPS to a randomized controlled trial in infancy (n=120), and among low-risk adolescents followed since middle childhood (n=80) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Must have been included in middle childhood data collection

Exclusion Criteria:

* None

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Brain activation in Stop Signal Task | Child age 13 years
  Prefrontal cortex activation assessed through functional magnetic resonance imaging (fMRI) in task requiring inhibitory control
Brain activation in Mother-Stranger Task | Age 13 years
  Functional connectivity assessed through fMRI when viewing photos of mothers vs. strangers
Brain activation in Mother-Stranger Task | Age 15 years
  Functional connectivity assessed through fMRI when viewing photos of mothers vs. strangers
Brain activation in Emotion Go/Nogo task | Age 13 years
  Functional connectivity between amygdala and PFC assessed through fMRI in an emotion go/no go task
Brain activation in Emotional Reappraisal Task | Age 14 years
  Functional connectivity between amygdala and PFC assessed through fMRI in emotional reappraisal task
Brain activation in Emotion Go/Nogo task | Age 15 years
  Functional connectivity between amygdala and PFC assessed through fMRI in an emotion go/no go task
Trier Social Stress Test- Cortisol | Age 13 years
  Participants will be met by two research assistants (one male, one female), whom they have not met previously. The research assistants will tell the participants that they will have 5 minutes to prepare a speech which they will give to the researchers who will rate the speech. Participants will then give their speeches for 5 minutes; the research assistants will maintain neutral expressions and provide no feedback. Afterwards, participants will be asked to do (age-adjusted) mental arithmetic aloud (Buske-Kirschbaum et al.,1997). For the purpose of assessing cortisol, investigators will collect saliva samples before and after the speech/math.
Trier Social Stress Test-ANS | Age 13 years
  Participants will be met by two research assistants (one male, one female), whom they have not met previously. The research assistants will tell the participants that they will have 5 minutes to prepare a speech which they will give to the researchers who will rate the speech. Participants will then give their speeches for 5 minutes; the research assistants will maintain neutral expressions and provide no feedback. Afterwards, participants will be asked to do (age-adjusted) mental arithmetic aloud (Buske-Kirschbaum et al.,1997).Assess child autonomic nervous system regulation, examine reactivity from baseline in RSA.
Revealed differences task - parent sensitivity. | Age 13 years
  Parents and children engage in conflict discussion. Assess parental sensitivity using Sensitivity scale. Parental behavior is scored on a 1-7 scale, with higher scores reflecting greater sensitivity.
Support task- parent sensitivity | Age 14 years
  Parents and children engage in support discussion (discussing Trier task from previous year). Assess parental sensitivity using Sensitivity scale. Parental behavior is scored on a 1-7 scale, with higher scores reflecting greater sensitivity.
Revealed differences task- parent sensitivity | Age 15 years
  Parents and children engage in conflict discussion. Assess parental sensitivity using Sensitivity scale. Parental behavior is scored on a 1-7 scale, with higher scores reflecting greater sensitivity.
Revealed differences task-adolescent competence | Age 13 years
  Parents and children engage in conflict discussion. Assess child competence in discussion on Competence scale. Competence is scored on a 1-7 scale, with higher scores reflecting greater competence.
Support task-adolescent competence | Age 14 years
  Parents and children engage in conflict discussion. Assess child competence in discussion on Competence scale. Competence is scored on a 1-7 scale, with higher scores reflecting greater competence.
Revealed differences task-adolescent competence | 15 years of age.
  Parents and children engage in conflict discussion. Assess child competence in discussion on Competence scale. Competence is scored on a 1-7 scale, with higher scores reflecting greater competence.
Revealed differences task-adolescent ANS | 13 years of age.
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout the parent-child interaction using a MindWare Portable Lab system. Greater changes in RSA from baseline to discussion considered preferable.
  Parents and children engage in conflict discussion. Assess child autonomic nervous system regulation. Respiratory sinus arrhythmia (RSA) will be measured as a rise from baseline.
Support task-adolescent ANS | 14 years of age.
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout the parent-child interaction using a MindWare Portable Lab system. Greater changes in RSA from baseline to discussion considered preferable.
Revealed differences task-adolescent ANS | 15 years of age.
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout the parent-child interaction using a MindWare Portable Lab system. Greater changes in RSA from baseline to discussion considered preferable.
Balloon Analogue Risk Task (BART) | 13 years of age
  This task assesses risk-taking through a computer game in which participants see a balloon on the computer screen and have the option of pumping up the balloon more, and therefore increasing its monetary value, or stopping and collecting the value of the balloon. If the balloon pops on a pump, then all of the value of the balloon is lost and the next trial begins. There is a randomly, pre-determined probability of the balloon popping on any given pump of each trial. A brief version of the task with 15 balloons will be used. A running tally of participants' total monetary gain is kept (and can range from $0 up to a cap of $5). The amount of money earned is the score, with more money reflecting higher risk taking.
Delay Discounting | 13 years of age
  Delay Discounting Task is a brief, five-item task on a computer that asks participants their preference between $5 now and $10 at some later time point (Koffarnus, Warren, & Bickel, 2014). No money is actually earned on this task. A score from 0 to 5 is received with lower score indicating better delay (preferred).
Delay Discounting | 15 years of age
  Delay Discounting Task is a brief, five-item task on a computer that asks participants their preference between $5 now and $10 at some later time point (Koffarnus, Warren, & Bickel, 2014). No money is actually earned on this task. A score from 0 to 5 is received with lower score indicating better delay (preferred).
Child Depression | 13 years of age
  Child Depression Inventory-Short Version (CDI-S): A 10-item measure that screens for depression (Kovacs, 2010). Scores can range from 0-24, with higher scores reflecting greater depression.
Child Depression | 14 years of age
  Child Depression Inventory-Short Version (CDI-S): A 10-item measure that screens for depression (Kovacs, 2010). Scores can range from 0-24, with higher scores reflecting greater depression.
Child Depression | 15 years of age
  Child Depression Inventory-Short Version (CDI-S): A 10-item measure that screens for depression (Kovacs, 2010). Scores can range from 0-24, with higher scores reflecting greater depression.
Child problem behaviors | 13 years of age
  Child Behavior Checklist (CBCL): Parents will complete the 113 items from the CBCL to assess adolescents' internalizing and externalizing symptoms (Achenbach et al., 2001). Raw scores range from 0-240. Higher scores reflect greater problems.
Child problem behaviors | 14 years of age
  Child Behavior Checklist (CBCL): Parents will complete the 113 items from the CBCL to assess adolescents' internalizing and externalizing symptoms (Achenbach et al., 2001). Raw scores range from 0-240. Higher scores reflect greater problems.
Child problem behaviors | 15 years of age
  Child Behavior Checklist (CBCL): Parents will complete the 113 items from the CBCL to assess adolescents' internalizing and externalizing symptoms (Achenbach et al., 2001). Raw scores range from 0-240. Higher scores reflect greater problems.
Adolescent substance use | 13 years of age
  Adolescents will complete the Youth Risk Behavior Survey. Higher scores reflect more substance use, with a possible range of 21-98.
Adolescent substance use | 14 years of age
  Adolescents will complete the Youth Risk Behavior Survey. Higher scores reflect more substance use, with a possible range of 21-98.
Adolescent substance use | 15 years of age
  Adolescents will complete the Youth Risk Behavior Survey. Higher scores reflect more substance use, with a possible range of 21-98.
Adolescent risky behaviors | 13 years of age
  Adolescents will complete the Youth Risk Behavior Survey. Higher scores reflect more risky problems, with a possible range of 8-28.
Adolescent risky behaviors | 14 years of age
  Adolescents will complete the Youth Risk Behavior Survey. Higher scores reflect more risky problems, with a possible range of 8-28.
Adolescent risky behaviors | 15 years of age
  Adolescents will complete the Youth Risk Behavior Survey. Higher scores reflect more risky problems, with a possible range of 8-28.
Mini-International Neuropsychiatric Interview for Children and Adolescents | 13 years of age
  Psychiatric interview. Higher scores reflect more psychiatric symptoms, with a range of 0-8.
Mini-International Neuropsychiatric Interview for Children and Adolescents | 14 years of age
  Psychiatric interview. Higher scores reflect more psychiatric symptoms, with a range of 0-8.
Emotional Regulation Questionnaire | 14 years of age
  Assesses how effectively adolescents regulate or control emotions. Higher scores reflect better regulation. Scores range from 10-50.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dozier, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
As described below, data will be made available to the scientific community for further analysis and novel research purposes after the primary results of the study have been published.
  De-identified research data will be shared in spreadsheet format for all clinical assessment, survey, and behavioral data. MRI data will be shared in NIFTI format. A description of the variables that are included in the dataset as well as a description of the data collection methods will also be provided. All data sharing will be done in consultation with our IRB.
  Results will be shared within one year of the completion of data collection of primary outcome measures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months following final data collection for at least 3 years.